CLINICAL TRIAL: NCT06641856
Title: Respiratory Virome Diversity and Baseline Immunity in Healthy Individuals in Shanghai
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, Professor, Ruijin Hospital
Other Study IDs: 202435
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Health Personnel
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Nasal and Pharyngeal Swabs: Two nasal swabs and three pharyngeal swabs will be collected from all 300 participants. These samples will be used for virome analysis to detect and characterize viruses present in the upper respiratory tract.
  2. Peripheral Blood: From a subset of 60 participants (30 young adults and 30 elderly individuals), 10 mL of peripheral blood will be drawn using sodium citrate anticoagulant tubes. The blood samples will be centrifuged to separate plasma and blood cells.
  3. Upper and Lower Respiratory Tract Samples: For the same subset of 60 participants, bronchoscopy will be performed under general anesthesia to collect respiratory tract samples from both the upper and lower airways.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Young Healthy Volunteers Group: Age Range: 20-35 years Health Status: Participants in this group must be in good overall health, as determined by medical history, physical examination, and results of a routine health check-up within the past year.
  Body Mass Index (BMI): Must be between 19-26 kg/m² (inclusive), with a minimum weight of 50 kg for males and 45 kg for females.
  Sample Size: 150 participants (including equal representation of males and females).
  Geographic Representation: Both permanent residents of Shanghai and non-residents who have been in the city for less than 30 days will be included. The proportion of local residents to non-residents will range from 1:1 to 2:1.
  Interventions: Other: Sample Collection
- Elderly Healthy Volunteers Group: Age Range: 60-75 years Health Status: Participants in this group must have good respiratory health and be generally healthy based on medical history, physical examination, and a health check-up within the past year.
  Body Mass Index (BMI): Must be between 19-26 kg/m² (inclusive), with a minimum weight of 50 kg for males and 45 kg for females.
  Sample Size: 150 participants (including equal representation of males and females).
  Geographic Representation: Similar to the young group, the elderly group will include both permanent residents of Shanghai and non-residents, with the same proportion of local residents to non-residents (1:1 to 2:1).
  Interventions: Other: Sample Collection

INTERVENTIONS:
Other: Sample Collection — All participants will provide nasal and pharyngeal swabs for virome analysis. A subset of 30 elderly volunteers will also provide peripheral blood samples and undergo bronchoscopy under general anesthesia to collect upper and lower respiratory tract samples.

SUMMARY:
This study investigates the diversity of the respiratory virome in healthy individuals in Shanghai and its interaction with the host's baseline immune response. The respiratory virome plays a critical role in various diseases, but research on the respiratory virome in healthy individuals in China is limited. This prospective study will analyze the upper and lower respiratory virome and examine the effects of demographic factors such as age, gender, and geographic background. Additionally, a respiratory virome database will be established, and multi-omics approaches will be used to study immune response mechanisms in relation to virome diversity.

DETAILED DESCRIPTION:
The study aims to provide comprehensive baseline data on the respiratory virome in healthy individuals in Shanghai. The primary goal is to investigate virome diversity in the upper and lower respiratory tracts and assess how demographic factors influence virome composition. Furthermore, the study will identify previously unknown viral sequences and explore their potential role in the immune system's interaction with the virome. Multi-omics approaches, including transcriptomics and proteomics, will be utilized to evaluate immune-related biomarkers and gene expression related to respiratory virome diversity.

ELIGIBILITY:
1. Young Healthy Volunteers

Inclusion Criteria:

1. Age between 20-35 years (inclusive), Han ethnicity, regardless of gender. Body Mass Index (BMI) between 19-26 kg/m² (inclusive), with a minimum weight of 50 kg for males and 45 kg for females.
2. The participant must be in good overall health, as determined by medical history, physical examination, vital signs, and results from a health checkup within the past year (normal or clinically insignificant findings).
3. Female participants must be non-pregnant and non-lactating.
4. Able to tolerate bronchoscopy and willing to provide nasal and pharyngeal swabs, as well as upper and lower respiratory secretions and peripheral blood samples.
5. Fully informed of the study's purpose, methods, and potential discomforts, with written informed consent provided, and willing to complete the study questionnaire.
6. Good compliance and willingness to follow the study protocol and complete follow-up procedures.

Exclusion Criteria:

1. Non-permanent residents of Shanghai who have stayed in the city for more than 30 days; or permanent residents of Shanghai who have left the city within the past 30 days.
2. History of significant illness or major surgery within the past 30 days, or anticipation of major surgery during the study period.
3. Diagnosis of respiratory diseases (infectious or non-infectious) within the past 30 days, requiring medication (oral, inhaled, or nebulized).
4. Presence of clinically significant diseases or factors, including but not limited to neurological, cardiovascular, hematologic, hepatic, renal, gastrointestinal, respiratory, metabolic, endocrine, immune, skeletal diseases, or other conditions deemed unsuitable by the investigator.
5. Long-term use of medication.
6. Positive test results for HIV antibodies (HIV-Ab), hepatitis B surface antigen (HBsAg), hepatitis C antibodies (HCV-Ab), or syphilis antibodies (TP-Ab).
7. Participation in any drug or medical device clinical trial within the past 3 months.
8. Vaccination within the past 30 days or planned vaccination during the study period.
9. Any other condition deemed by the investigator to impact the participant's ability to provide informed consent, follow the protocol, or affect study outcomes or the participant's safety.

2. Elderly Healthy Volunteers

Inclusion Criteria:

1. Age between 60-75 years (inclusive), Han ethnicity, regardless of gender. Body Mass Index (BMI) between 19-26 kg/m² (inclusive), with a minimum weight of 50 kg for males and 45 kg for females.
2. The participant must have a healthy respiratory system, as determined by medical history, physical examination, vital signs, and results from a health checkup within the past year (normal or clinically insignificant findings).
3. Able to tolerate bronchoscopy and willing to provide nasal and pharyngeal swabs, as well as upper and lower respiratory secretions and peripheral blood samples.
4. Fully informed of the study's purpose, methods, and potential discomforts, with written informed consent provided, and able to independently complete the study questionnaire.
5. Good compliance and willingness to follow the study protocol and complete follow-up procedures.

Exclusion Criteria:

1. Non-permanent residents of Shanghai who have stayed in the city for more than 30 days; or permanent residents of Shanghai who have left the city within the past 30 days.
2. History of significant illness or major surgery within the past 30 days, or anticipation of major surgery during the study period.
3. Diagnosis of respiratory diseases (infectious or non-infectious) within the past 30 days, requiring medication (oral, inhaled, or nebulized).
4. Presence of abnormal respiratory system function or other clinically significant diseases or conditions.
5. History of malignant tumors (including hematologic malignancies or solid tumors).
6. Long-term use of medication.
7. Positive test results for HIV antibodies (HIV-Ab), hepatitis B surface antigen (HBsAg), hepatitis C antibodies (HCV-Ab), or syphilis antibodies (TP-Ab).
8. Participation in any drug or medical device clinical trial within the past 3 months.
9. Vaccination within the past 30 days or planned vaccination during the study period.
10. Any other condition deemed by the investigator to impact the participant's ability to provide informed consent, follow the protocol, or affect study outcomes or the participant's safety.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include healthy Han Chinese individuals residing in Shanghai, divided into two age groups: young adults (20-35 years) and elderly individuals (60-75 years). A total of 300 participants will be recruited, regardless of gender. These participants will be selected based on good overall health, as determined by medical history, physical examination, and recent health checkup results.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Virome Composition and Diversity | From date of inclusion until the date of final quantification, assessed up to 6 months
  Characterization of respiratory virome diversity in upper and lower respiratory tracts of healthy individuals, measured through viral sequencing of nasal, throat, and bronchoscopic samples.
Host Immune Response | From date of inclusion until the date of final quantification, assessed up to 6 months
  Analysis of immune-related biomarkers and gene expression in blood samples, focusing on the interaction between respiratory virome diversity and the host immune response.

SECONDARY OUTCOMES:
Virome and Demographic Correlation | From date of inclusion until the date of final quantification, assessed up to 6 months
  Analysis of the correlation between virome composition and demographic factors such as age, gender, and geographic location.
Discovery of Unknown Viruses | From date of inclusion until the date of final quantification, assessed up to 6 months
  Identification of novel viral sequences and their potential immunological significance in healthy individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Jieming Qu, Ph. D, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No